CLINICAL TRIAL: NCT06573983
Title: Development of a Fall Risk Identification and Management Model for Older Veterans
Brief Title: Fall Risk Identification and Management for Older Veterans
Acronym: FRIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E5024-W
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Fall Risk
Keywords: Falls; Telerehabilitation; Multifactorial; Preventative; Personalized
MeSH Terms: interventions — Physical Therapy Modalities; Cognitive Behavioral Therapy; Psychology, Clinical; Occupational Therapy; Medication Reconciliation

STUDY DESIGN:
Intervention Model Description: There are two phases to the study. The first phase will include refinement of the intervention by examining quantitative and qualitative data from a small number of participants with no control. The second phase will be a randomized feasibility pilot where the intervention group will be compared to standard of care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors and investigators will be blinded to assignment during phase 2. Participants and care providers are unable to be blinded as delivery of treatment outside of standard of care will demonstrate group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fall Risk Identification and Management Model (Experimental): Participants will be assessed on four fall risk factors including physical, psychological, pharmacological, and environmental. If a participant screens positive for a fall risk factor, they will then be referred to an existing VHA care pathway. The care pathways include: strengthening via physical therapy or Gerofit for physical fall risk, cognitive behavioral therapy via clinical psychology or occupational therapy for psychological fall risk, deprescription via clinical pharmacy for pharmacological fall risk, and home safety modifications via occupational therapy for environmental fall risk.
  Interventions: Other: Strengthening (Physical Therapy, Gerofit); Other: Cognitive Behavioral Therapy (Clinical Psychology, Occupational Therapy); Other: Medication Reconciliation (Clinical Pharmacology); Other: Home Safety Modification (Occupational Therapy)
- Standard of care (No Intervention): This group will received current standard of care within the Rocky Mountain Regional GeriPACT clinic.

INTERVENTIONS:
Other: Strengthening (Physical Therapy, Gerofit) — Individuals with physical fall risk will be referred to strengthening interventions available within the VHA. These may include Physical Therapy or Gerofit (a supervised exercise program).
  Arms: Fall Risk Identification and Management Model
Other: Cognitive Behavioral Therapy (Clinical Psychology, Occupational Therapy) — Individuals with psychological fall risk will be referred psychological interventions such as cognitive behavioral therapy, which focuses on guided talking. This can be performed by VHA occupational therapists and clinical psychologists.
  Arms: Fall Risk Identification and Management Model
Other: Medication Reconciliation (Clinical Pharmacology) — Individuals with pharmacological fall risk will be referred to clinical pharmacology for medication reconciliation. This includes examining the current medication list and deprescribing medications, if appropriate.
  Arms: Fall Risk Identification and Management Model
Other: Home Safety Modification (Occupational Therapy) — Individuals with environmental fall risk will be referred to occupational therapy for home safety assessments and modifications. This will involve modifying components within the home to reduce potential fall risk factors.
  Arms: Fall Risk Identification and Management Model

SUMMARY:
Falls are a common occurrence among older adults, and Veterans have an even higher risk of falling compared to non-Veterans. These falls often lead to severe health consequences, including traumatic brain injuries, hip fractures, emergency visits, hospitalizations, and even death. It is crucial to prioritize fall prevention in order to reduce injuries and enable older Veterans to age comfortably at home. Although current fall prevention programs in the Veterans Health Administration primarily focus on inpatient care and nursing homes, there is a pressing need to address falls among older Veterans living independently in the community. The proposed VA-specific Fall Risk Identification and Management (FRIM) model aims to proactively prevent falls in older Veterans who receive primary care, effectively reducing the occurrence of adverse health events associated with falls. By placing emphasis on prevention rather than reacting after falls have already happened, this initiative seeks to significantly enhance the overall well-being of older Veterans.

DETAILED DESCRIPTION:
Falls among older adults pose a significant risk, leading to life-altering injuries and imposing substantial healthcare costs. There is a pressing need to develop fall prevention models within the Veterans Health Administration (VHA) considering Veterans are more likely to fall than their age-matched non-Veteran counterparts, likely secondary to higher rates of functional impairment and comorbidities. Extensive research has identified numerous fall risk factors across physical, psychological, pharmacological, and environmental domains. Further, screening tools and interventions have been developed to identify and manage these risk factors, offering insight on methods to intervene early and prevent falls in older Veterans. Primary care clinics within the VHA are well-positioned to play a crucial role in preventing falls. These clinics are frequently visited by older Veterans for routine care and are widely accessible across the country. However, fall risk assessment is often not included in the standard care provided by VHA primary care clinics, mainly due to barriers like limited time, competing medical priorities, and a lack of training. Consequently, there is a missed opportunity to address fall prevention. Therefore, the investigators are developing a personalized multifactorial model called Fall Risk Identification and Management (FRIM) to prevent falls in older Veterans seen within primary care by addressing known barriers that have limited the uptake of other fall prevention models. Specifically, the FRIM model follows a three-stage process: briefly screening for fall risk during routine primary care visits, conducting telehealth visits to identify specific fall risk factors, and referring Veterans to existing VHA care pathways with established interventions for managing identified risk factors. The objectives of this CDA-2 are to refine (Aim 1; Phase 1) and assess the feasibility (Aim 2; Phase 2) of the FRIM model in preparation for a future efficacy trial. The initial phase, Aim 1, focuses on refining the FRIM model by gathering feedback on each care pathway from Veterans and clinicians through qualitative interviews following a small field test. Additionally, the investigators will assess the impact of each care pathway on fall risk factor assessments. This phase aims to enhance the model based on the integration of perceptions and outcomes. Following the refinement of the FRIM model, Aim 2 entails conducting a randomized controlled feasibility pilot study. This phase will involve the collection of both qualitative and quantitative data to evaluate the feasibility, acceptability, and candidate efficacy outcomes of the FRIM model while comparing it to VHA standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Screens positive for increased fall risk within GeriPACT, or generalPACT as needed, (answers "yes" to any of 3 screening questions)
* 65 years of age and older
* Positive screen on at least two fall risk factor assessments (Aim 1); Positive screen on at least one fall risk factor assessment (Aim 2)
* Access to telehealth
* Availability of an additional adult (e.g., caregiver or family member) to be present during the physical assessment

Exclusion Criteria:

* Life expectancy <12 months, as determined by PCP
* Neurological diagnosis (e.g., cerebral vascular accident, multiple sclerosis, Parkinson's Disease)
* Moderate cognitive impairment (<13 on telephone Montreal Cognitive Assessment (MoCA-BLIND) or <18 on MoCA Full administered during clinic visit in the previous 3 months)
* Unstable condition that precludes safe participation in structured exercise (e.g., recent deep vein thrombosis) if expected fall risk factor is physical, as determined by PCP or chart review
* Participation in any intervention components of the FRIM model, with the intention of reducing a FRIM fall risk factor, within the past 2 months
* Currently using a wheelchair for mobilization
* If it is in the opinion of the study staff that the participant would be at an increased suicide risk due to study procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment | Program start
  Participant recruitment will be tracked as part of feasibility. It will be determined as the proportion of Veterans screened as eligible that are recruited.
Participant retention | Program start - 1 year post baseline
  Participant retention will be tracked as part of feasibility. It will be determined as the 1-year retention rate of participants.

SECONDARY OUTCOMES:
Fall risk identification burden | Program start, Program end (average of 12 weeks)
  Fall risk identification burden will be tracked as part of feasibility. It will be determined as the time to identify fall risk factors during telehealth visit.
Fall risk management burden | Program start - Program end (average of 12 weeks)
  Fall risk management burden will be tracked as part of feasibility. It will be determined as the time to complete fall risk factor management.
Theoretical framework of acceptability questionnaire | Program end (average of 12 weeks)
  Acceptability will be measured using an established questionnaire based on the theoretical framework of acceptability. Responses on the questionnaire range from 1 (did not like, high burden) to 5 (strongly liked, low burden).
3 key questions | Program start
  The 3 key questions include 1) whether the older adult feels unsteady when standing or walking, 2) worries about falling, 3) or has fallen in the past year. Participant responses of 'yes' or 'no' to each question will be recorded.
5 times sit to stand | Program start, 1 year after intervention end (average of 1.25 years post baseline)
  The 5 times sit to stand is a test of lower extremity strength, transitional movements, and balance. The test is scored based on the time to completed 5 sit to stand movements and is highly predictive of falls and injurious falls. A higher time indicates worse physical function and greater physical fall risk.
Survey of Activities and Fear of Falling in the Elderly | Program start, 1 year after intervention end (average of 1.25 years post baseline)
  This survey is a questionnaire that probes fear of falling and activity restriction of eleven activities. Fear of falling is scored based on the average worry to perform each activity ranging from 0 (not worried) to 3 (very worried). Activity restriction is scored by the number of activities that an individuals reports doing less than usual compared to three years ago. Additional questions probe whether activities are restricted due to fear of falling. Higher scores indicate greater psychological fall risk.
Screening Tool of Older Persons Prescriptions in older adults with high fall risk (STOPPFall) | Program start, 1 year after intervention end (average of 1.25 years post baseline)
  Pharmacological fall risk will be identified via the number of medications prescribed on the Screening Tool of Older Persons Prescriptions in older adults with high fall risk. The number of medications prescribed will be collected from the participant's medical record. A higher score indicates more fall risk increasing drugs and greater pharmacological fall risk.
Home Falls and Accidents Screening Tool (HOME FAST) | Program start, 1 year after intervention end (average of 1.25 years post baseline)
  The Home Falls and Accidents and Screening Tool is a questionnaire that assesses 25 potential home fall risk factors (e.g., slippery surfaces, lighting, etc.). A higher score indicates greater environmental fall risk.
Unique number of falls. | Through study completion (average of 1.25 years)
  Unique number of falls will be measured as a yes/no occurrence of any falls during the study. This will be measured using weekly self-report via the Annie-App as well as using the VA Data Corporate Warehouse.
Median cumulative number of falls | Through study completion (average of 1.25 years)
  Median number of cumulative falls per Veteran will be collected using weekly self-report via the Annie-App as well as using the VA Data Corporate Warehouse.
Time to first fall | Through study completion (average of 1.25 years)
  Time to first fall is a continuous measure of days to the first fall occurring within the study period. This will be collected using weekly self-report via the Annie-App as well as using the VA Data Corporate Warehouse.
Unique number of injurious falls | Through study completion (average of 1.25 years)
  Injurious falls will be defined as falls requiring medical attention. Unique number of injurious falls will be measured as a yes/no occurrence of any injurious falls during the study. This will be measured using weekly self-report via the Annie-App as well as using the VA Data Corporate Warehouse.
Median cumulative number of injurious falls | Through study completion (average of 1.25 years)
  Injurious falls will be defined as falls requiring medical attention. Median number of cumulative injurious falls per Veteran will be collected using weekly self-report via the Annie-App as well as using the VA Data Corporate Warehouse.
Time to first injurious fall | Through study completion (average of 1.25 years)
  Injurious falls will be defined as falls requiring medical attention. Time to first injurious fall is a continuous measure of days to the first injurious fall occurring within the study period. This will be collected using weekly self-report via the Annie-App as well as using the VA Data Corporate Warehouse.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Garbin, PhD DPT, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team intends to share study data that may be requested from other research investigators in a data-sharing agreement provided at the study's end. Data prepared for distribution under a data-sharing agreement will be further redacted to ensure privacy of study participant identity yet allow analyses to occur by other investigators. The data-sharing agreement will include requirements to protect participants' privacy and data confidentiality.
Time Frame: 6 months after publication
Access Criteria: The research team intends to share study data that may be requested from other research investigators in a data-sharing agreement provided at the study's end.